CLINICAL TRIAL: NCT07308613
Title: Developing and Testing a Machine Learning Enabled Mindfulness Intervention for Reducing Loneliness Among Hong Kong Chinese Older Adults: A Hybrid Experimental Design Study
Brief Title: Developing and Testing a Machine Learning Enabled Mindfulness Intervention for Reducing Loneliness Among Hong Kong Chinese Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Chou Kee Lee, Chair Professor, Education University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-2024-0147
Record Dates: First submitted 2025-12-08; First posted 2025-12-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Loneliness
Keywords: Loneliness; Older Adults; Mindfulness; hybrid SMART-MRT

STUDY DESIGN:
Intervention Model Description: A hybrid factorial-SMART-MRT experimental design with a 2x2+1 factorial design (with five arms) randomized clinical trial, a two-stage SMART, and three MRTs will be utilized.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- App & Human Coaching + Continue Intervention (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (App + Human Coaching) Responder
  Interventions: Behavioral: Mindfulness - Continue
- Active Control (Active Comparator): Active Control
  Interventions: Behavioral: Active Control
- App & Human Coaching + Increase intensity in human coaching (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (App + Human Coaching) Non-Responder
  Interventions: Behavioral: Mindfulness - Enhance human coaching
- App & Human Coaching + Booster (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (App + Human Coaching) Non-Responder
  Interventions: Behavioral: Mindfulness - Booster
- App Coaching + Continue Intervention (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (App Coaching) Responder
  Interventions: Behavioral: Mindfulness - Continue
- App Coaching + Increase intensity in human coaching (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (App Coaching) Non-Responder
  Interventions: Behavioral: Mindfulness - Enhance human coaching
- App Coaching + Booster (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (App Coaching) Non-Responder
  Interventions: Behavioral: Mindfulness - Booster
- Human Coaching + Continue Intervention (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (Human Coaching) Responder
  Interventions: Behavioral: Mindfulness - Continue
- Human Coaching + Increase intensity in human coaching (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (Human Coaching) Non-Responder
  Interventions: Behavioral: Mindfulness - Enhance human coaching
- Human Coaching + Booster (Experimental): First-line of coaching (4 weeks):
  Single-Session Intervention of Mindfulness (Human Coaching) Non-Responder
  Interventions: Behavioral: Mindfulness - Booster
- No Coaching + Continue Intervention (Experimental): First-line of coaching (4 weeks):
  No Single-Session Intervention of Mindfulness Responder
  Interventions: Behavioral: Mindfulness - Continue
- No Coaching + Increase intensity in human coaching (Experimental): First-line of coaching (4 weeks):
  No Single-Session Intervention of Mindfulness Non-Responder
  Interventions: Behavioral: Mindfulness - Enhance human coaching
- No Coaching + Booster (Experimental): First-line of coaching (4 weeks):
  No Single-Session Intervention of Mindfulness Non-Responder
  Interventions: Behavioral: Mindfulness - Booster

INTERVENTIONS:
Behavioral: Mindfulness - Continue — Second-line of coaching (4 weeks):
  Continue with existing intervention plan
  Arms: App & Human Coaching + Continue Intervention; App Coaching + Continue Intervention; Human Coaching + Continue Intervention; No Coaching + Continue Intervention
Behavioral: Mindfulness - Enhance human coaching — Second-line of coaching (4 weeks):
  Increase intensity of human coaching
  Arms: App & Human Coaching + Increase intensity in human coaching; App Coaching + Increase intensity in human coaching; Human Coaching + Increase intensity in human coaching; No Coaching + Increase intensity in human coaching
Behavioral: Mindfulness - Booster — Second-line of coaching (4 weeks):
  Add a booster session
  Arms: App & Human Coaching + Booster; App Coaching + Booster; Human Coaching + Booster; No Coaching + Booster
Behavioral: Active Control — No rerandomization, no mindfulness, No MRT
  Arms: Active Control

SUMMARY:
Develop and test an effective machine learning enabled application-based (app-based) mindfulness intervention for reducing loneliness of Hong Kong Chinese older adults.

DETAILED DESCRIPTION:
This study will utilize a hybrid Sequential Multiple Assignment Randomized Trial-Micro Randomized Trial (Hybrid SMART-MRT) to: 1) evaluate the effectiveness of a single-session intervention (SSI) of mindfulness on reducing loneliness; 2) identify the optimal first-line coaching approach after the SSI of mindfulness; 3) examine whether increasing the intensity of human coaching or adding a telephone-based human-delivered booster session will benefit participants who do not respond to the first-line coaching; 4) determine whether sending push notifications increases the engagement of our app-based coaching, by comparing its results with those of no push notification; 5) determine whether sending a recommended activity increases the engagement of our app-based coaching, by comparing its results with those of no recommended activity; and 6) determine whether sending a personalized motivational message increases the engagement of our app-based coaching, by comparing its results with those of a standard motivational message.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older
* Possess a smartphone with an Android or iOS operating system
* Communicable in Cantonese
* Lonely (cut-off >/=6 on the three-item UCLA Loneliness Scale)

Exclusion Criteria:

* Cognitive impairment, psychiatric disorder, learning disability
* Active suicide ideation
* Engaged in psychotherapy and psychosocial interventions in the past year

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  UCLA Loneliness Scale; each item will be rated from 1=Never to 4=Always. Total scores range from 20 to 80

SECONDARY OUTCOMES:
Loneliness | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  De Jong Gierveld Loneliness Scale; each item will be rated from 1=Yes to 3=No. Total scores range from 0 to 6, with subscale score ranging from 0 to 3.
Stress | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Perceived Stress Scale; each item will be rated from 0=Never to 4=Very often. Total scores range from 0 to 56.
Sleep Quality | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Pittsburgh Sleep Quality Index; each item will be rated from 0=No difficulty to 3=Severe difficulty. Total scores range from 0 to 21.
Depression | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Patient Health Questionnaire-9; Each item will be rated from 0=Not at all to 3=nearly everyday. Total scores range from 0 to 27
Anxiety | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Generalised Anxiety Disorder; each item will be rated from 0=not at all to 3=nearly every day. Total score range from 0 to 21.
Physical Health | Baseline (T0), 6 months after 2nd-line of coaching (T4)
  Lawton Instrumental Activities of Daily Living; each item will be rated 0=dependent to 1=independent. Total scores range from 0 to 8.
Physical Health | Baseline (T0), 6 months after 2nd-line of coaching (T4)
  Activities of Daily Living; each item will be rate from 0=dependent to 5/10=independent. Total scores range from 0 to 100.
Physical Symptoms | Baseline (T0), 6 months after 2nd-line of coaching (T4)
  Wahler Physical Symptoms Inventory; each item will be rated from 0=almost never agree to 5=agree almost every day. Total score range from 0 to 210.
Chronic Illness | Baseline (T0), 6 months after 2nd-line of coaching (T4)
  Participants will indicate any presence of chronic illness (e.g., diabetes, asthma, high blood pressure).
Multidimensional Scale of Perceived Social Support | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  MSPSS evaluates the social support derived from three key sources: family, friends, and significant others. Each item will be rated from 1=Strongly disagree to 7=Strongly agree. Total scores range from 12 to 84.
Lubben Social Network Scale | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  LSNS is used to assess the social networks of participants. Each item will be rated 0=None to 5=9 or more. Total scores range from 0 to 30.

OTHER OUTCOMES:
Mindfulness | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Mindfulness Attention Awareness Scale; each item will be rated from 1=Almost always to 6=Almost never. Average score will be calculated.
Perceived Social Support | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Each item is rated on a 7-point Likert scale ranging from 1=Strongly disagree to 7=Strongly agree. Total scores range from 12 to 84, with subscale score ranging from 4 to 28. A higher score indicates higher levels of perceived support.
Social Isolation | Baseline (T0), within 1 week after 1st-line of coaching (T1), within 1 week after 2nd-line of coaching (T2), 3 months after 2nd-line of coaching (T3), 6 months after 2nd-line of coaching (T4)
  Lubben Social Network Scale; Each item is rated on a 6-point Likert scale ranging from 0=None to 5=9 or more. Total scores range from 0 to 30, with a higher score indicating greater social engagement and lower risk of social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Kee Lee Chou, PhD, Principal Investigator — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be available upon reasonable request.